CLINICAL TRIAL: NCT01165645
Title: Lopinavir/Ritonavir as an Immunomodulator to Enhance Vaccine Responsiveness
Brief Title: Lopinavir and Ritonavir in Improving Immune Response to Vaccines in Patients With Complete Remission Following A Bone Marrow Transplant for Hodgkin Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1083; NCI-2010-00880 (Registry Identifier: NCI's CTRO); MC1083 (Other: Mayo Clinic Cancer Center); 08-006246 (Other: Mayo Clinic IRB); 21096 (Other: Abbott Lab Protocol)
Record Dates: First submitted 2010-07-14; First posted 2010-07-20 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2015-10

CONDITIONS: Hodgkin Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage IV Adult Hodgkin Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Lopinavir; Ritonavir; Polymerase Chain Reaction; Flow Cytometry; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral lopinavir and ritonavir twice daily for 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lopinavir; Drug: ritonavir; Genetic: polymerase chain reaction; Other: flow cytometry; Other: enzyme-linked immunosorbent assay; Other: laboratory biomarker analysis
- Arm II (No Intervention): Patients receive no therapy.

INTERVENTIONS:
Drug: lopinavir — Given orally
  Other Names: ABT-378/r
  Arms: Arm I
Drug: ritonavir — Given orally
  Other Names: Norvir; RIT
  Arms: Arm I
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
  Arms: Arm I
Other: flow cytometry — Correlative studies
  Arms: Arm I
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
  Arms: Arm I
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I

SUMMARY:
RATIONALE: HIV protease inhibitors, including Lopinavir/Ritonavir have intrinsic anti-apoptotic properties in addition to their anti-viral effect on HIV. This anti-apoptotic effect may boost the immune system to help the body create a better immune response to vaccines. PURPOSE: This randomized clinical trial studies giving lopinavir and ritonavir together in improving immune response to vaccines in patients with complete remission following a bone marrow transplant for Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Compare TREC positive recent thymic emigrants, and naive CD4+ and CD8+ T cell numbers between treatment groups. SECONDARY OBJECTIVES: I. Compare post-vaccination anti-rabies antibody titers between treatment groups. II. Compare post-vaccination cytokine levels, including IL1, IL2, IL4, IL6, IL7, IL8, IL10, IL12, INFgamma, TNFalpha, between treatment groups. III. Compare post-vaccination anti-rabies ELISPOT reaction between treatment groups. OUTLINE: Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive oral lopinavir and oral ritonavir twice daily for 28 days in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive no therapy. All patients then receive a neo-antigen rabies vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects who are in complete remission at Day +100 after a bone marrow transplant for Hodgkins Lymphoma
* Normal AST or ALT, serum creatinine and 12-lead electrocardiogram within the previous 6 months
* Females of childbearing potential must have negative beta-HCG (urine or plasma) within the last month and agree to effective contraception during the course of the study
* Willingness and ability to give informed consent
* Willingness and ability to take pills twice a day for 28 days

Exclusion Criteria:

* Known HIV positive
* Screening ALT or AST greater than 3X upper limit of normal
* Baseline QTc greater than 500 msec
* Current treatment with immunosuppressive agent (systemic glucocorticoid, cyclosporine, mycophenolate, azathioprine, sirolimus, Rituximab, infliximab, adalimumab)
* Current treatment with any of the following: cisapride, ergot derivatives, amiodarone, quinidine, terfenadine, astemizole, rifampin/rifabutin, carbamazepine, phenobarbital, sildenafil, St. John's wort, azithromycin, carbamazepine, HIV anti-virals, methadone, pimozide, phenytoin, sedative hypnotics (midazolam, triazolam), HMG-CoA reductase inhibitors (lovastatin, simvastatin, atorvastatin)
* Active malignancy requiring chemotherapy or radiation
* Baseline creatinine of > 2.0
* Active infection requiring systemic anti-infective agent (excluding prophylactic antibiotics)
* Hypersensitivity to processed bovine gelatin, chicken protein, neomycin, amphotericin B or chlortetracycline
* Subject must not be on medications that interact with the metabolism of protease inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-12-14 (Actual)

PRIMARY OUTCOMES:
Comparison of TREC positive recent thymic emigrants, and naive CD4+ and CD8+ T cell numbers between treatment groups | 90 days

SECONDARY OUTCOMES:
Comparison of post-vaccination anti-rabies antibody titers between treatment groups | 90 days
Comparison of post-vaccination cytokine levels, including IL1, IL2, IL4, IL6, IL7, IL8, IL10, IL12, INFgamma, TNFalpha, between treatment groups | 90 days
Comparison of post-vaccination anti-rabies ELISPOT reaction between treatment groups | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Rizza, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States